CLINICAL TRIAL: NCT06949579
Title: Risk of Posterior Staphyloma in Highly Myopic Europeans : From Epidemiology to Anatomy.
Acronym: MYOFORTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP240842
Record Dates: First submitted 2025-03-24; First posted 2025-04-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: High Myopia
Keywords: High myopia; Myopic staphyloma
MeSH Terms: interventions — Blood Specimen Collection; DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AM A : High Myopia without myopic staphyloma (Experimental)
  Interventions: Biological: blood sampling for DNA
- ARM B : High myopia with myopic staphyloma (Active Comparator)
  Interventions: Biological: blood sampling for DNA

INTERVENTIONS:
Biological: blood sampling for DNA — Blood sampling for DNA and serum and plasma colection and PBMC

SUMMARY:
In this cross-sectionnal study the aim is to increase the understanding of posterior staphyloma through a unique European consortium. Therefore, all eligible patients that either visit the outpatient clinic at Radboud in Nimegen, the Netherlands, or visit University Hopital Puerta de HierroMajadahonda in Madrid, Spain, or visit University Hospital Cochin in Paris, France, and after consenting, will be included.

600 high myopic European cases are expecting. A standardized protocol in all centers in order to create a uniform dataset.

Besides the standard of care, blood samples will be collected.

All data collected will be stored in an onlie Castor database

DETAILED DESCRIPTION:
Main objective: To characterize the phenotype, genetics and biology of myopic staphyloma in a European population (three countries involved).

Primary Outcome Measure:

The primary objective of this study is to identify genetic variants (SNPs) significantly associated with the presence of posterior staphyloma in individuals of European ancestry with high myopia.

A genome-wide association study (GWAS) will be conducted in 600 highly myopic Caucasian participants, divided into two well-phenotyped groups:

* 300 patients with posterior staphyloma (case group)
* 300 patients without posterior staphyloma (control group) SNP allele frequencies will be compared between the two groups using logistic regression models adjusted for relevant covariates (age, sex, axial length, and genetic ancestry via principal components).

The primary endpoint is the identification of SNPs s reaching genome wide significance (p < 5×10-⁸)after correction for multiple testing.

Secondary Outcome Measures:

1. Functional annotation and biological pathway enrichment of associated loci Genome-wide significant SNPs will undergo functional annotation to identify nearby genes, regulatory regions, or non-coding variants with putative biological function.

   Pathway and gene ontology enrichment analyses (e.g., KEGG, Reactome, GO) will be performed to highlight potential biological mechanisms contributing to posterior staphyloma pathogenesis.
2. Association with retinal imaging phenotypes Exploratory analyses will assess the relationship between genome wide significant variants and quantitative retinal imaging traits, including: subfoveal choroidal thickness,axial length,staphyloma depth, stpahyloma location, scleral curvature… These associations will be evaluated using multivariable linear regression models, adjusted for potential confounders.
3. Association with structural complications of posterior staphyloma Further exploratory analyses will investigate whether genome wide significant

   SNPs are associated with major strutural complications of posterier staphyloma, such as :

   macular atrophy,Bruch's membrane ruptures,choroidal neovascularization,foveoschisis, retinal detachment, visual fonction These analyses aim to uncover genetic markers linked to disease severity or progression
4. Differential expression of disease-relevant plasma/ serum protein biomarkers between groups, quantified by mass spectrometry, and correlated with clinical phenotype severity or progression (e.g., visual acuity loss, anatomical changes on OCT)
5. Efficiency and quality of iPSC reprogramming from peripheral blood mononuclear cells (PBMCs) in each study group, 4 individuals (1 male and 1 female myopic patient with staphyloma and 1 male and 1 female myopic patient without staphyloma, aged 30 to 35) assessed by reprogramming success rate, pluripotency marker expression, and genomic integrity. Derived iPSCs will be used differentiate retinal pigment epithelial cells in order to compare disease-relevant cellular phenotypes and functional responses in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Adults with high myopia (axial length ≥ 26.00 mm or degree of myopia of at least -6 diopters), with and without posterior staphyloma

  * Adults aged 18 years or over
  * Patient with high myopia (axial length ≥ 26.00 mm or degree of myopia of at least -6 diopters), with good quality retinal imaging
  * Patient who has signed a consent form to participate in the study
  * Patient who is a beneficiary of a social security scheme or who is entitled to it

Exclusion Criteria:

* Any systemic or ocular pathologies with an impact on the posterior segment of the eye

  * Patient with a systemic pathology likely to affect the posterior segment of the eye:
  * Diabetes
  * Systemic inflammatory disease: sarcoidosis, rheumatoid arthritis, systemic lupus erythematosus, Horton's disease
  * Patients with retinitis pigmentosa
  * Patients with syndromic myopia
  * Patients with myopia associated with a genetic disease such as hereditary vitreoretinopathy
  * Patients under guardianship, curatorship or legal protection, as well as pregnant or breastfeeding women (article L1121-5 of the CSP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Differential gene expression between myopic patients with and without staphyloma | Through study completion, an average of 1 year.
  Genetic analysis

SECONDARY OUTCOMES:
Establish correlations between the phenotype and systemic molecular markers | Through study completion, an average of 1 year.
  Proteomic analysis in blood
Compare phenotype of staphyloma between France and 2 other European countries: Netherlands and Spain | 25 months
  Retinal imaging

CONTACTS AND LOCATIONS:
Overall Officials: Francine BEHAR-COHEN, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No